CLINICAL TRIAL: NCT07185737
Title: Cultural Adaptation of Parent Training Intervention for Spanish-Speaking Families
Brief Title: Culturally Adapted RUBI-T for Spanish-Speaking Families in Texas and Mexico
Acronym: SS RUBI-T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: University of Texas Rio Grande Valley (Other)
Responsible Party: Principal Investigator, Gospel Kim, Assistant Professor, Baylor University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2297844-2
Record Dates: First submitted 2025-09-13; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Autism
Keywords: Autism; Cultural Adaptation; RUBI-T; Behavior Parent Training
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two arms: (1) intervention arm, where caregivers immediately receive the culturally adapted RUBI program, or (2) waitlist control arm, where caregivers receive the same intervention after the first group completes the program.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted RUBI-T (Experimental): Caregivers randomized to this arm will immediately participate in the culturally adapted Research Units in Behavioral Intervention (RUBI) program. The intervention consists of 8 weekly group sessions delivered virtually in Spanish by trained behavioral therapists. Caregivers will also use a Spanish-language RUBI parent handbook to complete home practice assignments and will receive guided feedback and coaching during sessions.
  Interventions: Behavioral: Adapted RUBI-Telehealth
- Waitlist Control Arm (No Intervention): Spanish-speaking caregivers are placed on a waitlist and continue with usual care during the initial study period. After the intervention group completes the program, waitlist participants receive the same adapted RUBI program (8 weekly online sessions).

INTERVENTIONS:
Behavioral: Adapted RUBI-Telehealth — The Adapted RUBI Parent Training is a culturally tailored version of the Research Units in Behavioral Intervention (RUBI) program, designed for Spanish-speaking caregivers of young autistic children. The intervention consists of 8 weekly sessions delivered virtually in Spanish by trained behavioral therapists. Each session incorporates behavioral skills training methods (instruction, modeling, role-play, and feedback). Caregivers use a Spanish-language RUBI handbook to complete weekly home practice activities and receive feedback during sessions. The program focuses on helping caregivers understand the functions of challenging behavior and apply evidence-based strategies to reduce these behaviors and promote positive child outcomes.
  Arms: Adapted RUBI-T

SUMMARY:
Supporting young autistic children can sometimes be very stressful, especially when children show behaviors that are difficult to understand and/or manage in everyday life. Research has shown that teaching parents practical strategies through programs like the Research Units in Behavioral Intervention (RUBI) can reduce these behaviors and help parents feel more confident. However, most of these programs have only been studied with English-speaking families, which means Spanish-speaking caregivers often do not have access to support that feels relevant to their culture and language.

This study will test a version of RUBI that has been adapted for Spanish-speaking families in the U.S. and Mexico. We will invite 100 parents of autistic children between the ages of 2 and 9 to take part. Half will start the program right away, while the other half will wait and receive it later. Parents in the program will join eight online group sessions, use a Spanish handbook at home, and practice strategies with support from trained facilitators.

We will look at whether the program helps reduce children's challenging behaviors, lowers parent stress, and increases parents' confidence in managing behaviors. We will also ask parents to share their experiences and opinions about how well the program fits their culture and daily life.

By combining numbers (surveys) and stories (interviews), this project will show whether the adapted program works well for Spanish-speaking families. The results can help make autism services more fair, accessible, and supportive for families from diverse backgrounds.

DETAILED DESCRIPTION:
Background and Rationale Challenging behaviors in young autistic children can negatively affect their quality of life and increase stress for caregivers. Behavioral Parent Training (BPT) programs, such as the Research Units in Behavioral Intervention (RUBI), have demonstrated strong evidence for reducing child behavior difficulties and improving parenting outcomes. However, most studies have been conducted with White, English-speaking families, limiting generalizability to diverse communities. Spanish-speaking families in the United States and Mexico often experience limited access to culturally responsive interventions, creating disparities in autism care.

Cultural adaptation is a systematic approach to tailoring interventions to better align with the values, language, and lived experiences of target populations. Research indicates that culturally adapted interventions can improve both child and caregiver outcomes, but adaptation practices are inconsistently reported. Adapting RUBI for Spanish-speaking caregivers has the potential to increase its accessibility and effectiveness for an underserved group.

Objectives

This study aims to evaluate the effectiveness, feasibility, and cultural acceptability of an adapted RUBI program for Spanish-speaking caregivers of autistic children. The specific objectives are to:

1. Determine whether the adapted program reduces children's challenging behaviors.
2. Assess changes in caregiver stress, confidence, and knowledge of behavior strategies.
3. Examine caregiver perceptions of cultural relevance and satisfaction with the program.
4. Identify barriers and facilitators to program implementation.

Study Design This study uses a convergent mixed-methods design combining a pilot randomized controlled trial (RCT) with qualitative data collection. A total of 100 caregivers will be randomly assigned to either (a) the immediate intervention group or (b) the waitlist control group, who will receive the intervention after the initial study period.

Participants and Recruitment Caregivers will be recruited through community organizations, autism advocacy groups, ABA clinics, and online platforms serving Spanish-speaking families. Eligible participants must (a) be a caregiver of a child aged 2-9 years diagnosed with or suspected of autism, (b) report child challenging behaviors in everyday settings, (c) be Spanish-speaking, and (d) have access to internet and a device for online participation. Exclusion criteria include prior experience with RUBI.

Recruitment, consent, and baseline data collection will occur online. Participants will be enrolled beginning September 2025, with intervention delivery from September-November 2025 (intervention group) and January-March 2026 (waitlist control).

Intervention

The intervention is an eight-session, virtually delivered version of RUBI, culturally adapted for Spanish-speaking families. Parents will:

(a) Attend weekly group sessions via Zoom led by trained behavioral therapists; (b) Use a Spanish-language RUBI handbook for guided practice at home; (c) Engage in role-play, modeling, and practice with feedback based on behavioral skills training.

Outcomes Quantitative measures will include: (a) RUBI Parent Confidence Scale (PCS), (b) Home Situations Questionnaire-ASD (HSQ-ASD), (c) Caregiver Knowledge Assessment (CKA), (d) Scale of Treatment Perceptions (STP), (e) Autism Parent Stress Index (APSI), and (f) Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM).

Qualitative data will be collected through post-intervention open-ended responses and optional focus groups in Spanish, focusing on feasibility, satisfaction, and cultural relevance.

Analysis Plan Quantitative data will be analyzed using repeated measures ANOVA with time (pre vs. post) as a within-subject factor and condition (intervention vs. control) as a between-subject factor. Post hoc tests and Cohen's d will estimate effect sizes. Qualitative data will undergo rapid analysis by bilingual coders to identify themes related to program benefits, cultural fit, and implementation barriers. Triangulation across survey, focus group, and observational data will be used to strengthen findings.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of a child aged 2 to 9 years.
* Caregiver of a child diagnosed with autism or suspected of being autistic.
* Child exhibits challenging behaviors in naturalistic environments (e.g., home, school, community).
* Caregiver is willing to complete all aspects of the study, including assessments and intervention sessions.
* Caregiver has access to electronic resources (e.g., high-speed internet and a device capable of participating in Zoom sessions).
* Caregiver is fluent in Spanish (speaks and understands Spanish sufficiently to participate in the intervention and assessments).

Exclusion Criteria:

* Prior participation in the Research Units in Behavioral Intervention (RUBI) program.
* Caregiver does not speak Spanish.
* Caregiver unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in challenging behaviors measured by the Home Situations Questionnaire-ASD (HSQ-ASD) | Baseline (T1, pre-intervention), Post-intervention (T2, ~8 weeks after baseline), and Maintenance (T3, ~16 weeks after baseline, following waitlist group intervention)
  The HSQ-ASD (Chowdhury et al., 2016) is a 24-item caregiver-report tool assessing severity of challenging behaviors in children with autism across daily situations. Higher scores indicate more severe problem behaviors.
Change in caregiver confidence measured by the RUBI Parent Confidence Scale (PCS) | T1 (baseline), T2 (~8 weeks), and T3 (~16 weeks)
  The PCS is a 12-item measure of caregiver confidence in applying behavioral strategies from the RUBI program. Scores range from 1-3, with higher scores indicating greater confidence.
Change in caregiver knowledge measured by the Caregiver Knowledge Assessment (CKA) | T1 (baseline), T2 (~8 weeks), and T3 (~16 weeks)
  The CKA (Lee et al., 2022) is a 28-item multiple-choice assessment of caregiver knowledge of behavioral parent training strategies. Higher scores reflect greater knowledge.
Change in treatment acceptability and satisfaction measured by the Scale of Treatment Perceptions (STP) | T1 (baseline, anticipated outcomes), T2 (~8 weeks, satisfaction), and T3 (~16 weeks, maintenance satisfaction)
  The STP (Berger et al., 2016) uses a 7-point Likert scale to assess acceptability, anticipated outcomes (T1), and satisfaction with the program (T2, T3).

SECONDARY OUTCOMES:
Change in caregiver stress measured by the Autism Parenting Stress Index (APSI) | T1 (baseline, pre-intervention), T2 (post-intervention, ~8 weeks), and T3 (maintenance, ~16 weeks after baseline, following waitlist intervention)
  The APSI is a caregiver-report questionnaire that measures stress related to parenting a child with autism, focusing on areas such as social communication, challenging behaviors, and daily care. Higher scores indicate higher parenting stress.
Implementation outcomes of adapted RUBI program (12-item measure) | T3 (maintenance, ~16 weeks after baseline, following waitlist intervention)
  A 12-item implementation outcome measure will be used to assess caregiver perceptions of feasibility, acceptability, appropriateness, and intention to use the strategies taught in the adapted RUBI program. Items are scored on a Likert scale, with higher scores reflecting more favorable implementation outcomes.

OTHER OUTCOMES:
Caregiver perceptions of cultural relevance, feasibility, and barriers to implementation | Post-intervention (T2, ~8 weeks) and Maintenance (T3, ~16 weeks)
  Qualitative data will be collected through post-intervention narrative responses and optional semi-structured focus group interviews. Analyses will explore caregivers' experiences with cultural relevance, feasibility, barriers, and facilitators of the adapted RUBI program.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
The research team has not yet determined whether de-identified individual participant data (IPD) will be shared. Decisions will depend on IRB guidance, funding agency requirements, and feasibility of preparing anonymized datasets while maintaining participant confidentiality.